CLINICAL TRIAL: NCT05792267
Title: Clinical Research on Navigation and Quality Control System of Pancreatic Ultrasound Endoscopy Based on Deep Learning
Brief Title: Clinical Research on a Novel Deep-learning Based System in Pancreatic Endoscopic Ultrasound Scanning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-EUS-AI-001
Record Dates: First submitted 2023-03-17; First posted 2023-03-31 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Disease
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-assisted group (Experimental): Subjects will undergo EUS examination with the assistance of artificial intelligence(AI) system.
  Interventions: Device: artificial intelligence system
- Non-assisted group (No Intervention): Subjects will undergo EUS examination without the assistance of artificial intelligence(AI) system.

INTERVENTIONS:
Device: artificial intelligence system — Patients will undergo EUS examination with the assistance of artificial intelligence(AI) system.
  Arms: AI-assisted group

SUMMARY:
The goal of this clinical trial is to develop and verify the auxiliary role of the artificial intelligence system in pancreatic ultrasound endoscopic scanning.The main questions it aims to answer are as follows: 1.The comparison of the image recognition accuracy between the artificial intelligence system and the ultrasound endoscopist; 2. Whether the artificial intelligence system can improve the efficiency of the pancreatic scanning for the ultrasound endoscopist. Participants will undergo pancreatic EUS with or without the assistance of the artificial intelligence system.

DETAILED DESCRIPTION:
In this study, pancreatic endoscopic ultrasound scanning videos and images will be collected. First of all, an artificial intelligence system based on deep learning for the navigation and quality control of pancreatic endoscopic ultrasonography will be established. Secondly, the artificial intelligence system will be used to identify the site and anatomical structure of the pancreatic ultrasound endoscopy, and the results of the artificial intelligence system's station recognition will be compared with the results of the endoscopist's station recognition. Finally, the completeness of standard sites and scanning time of endoscopic-assisted and non-assisted AI systems were compared.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old, <80 years old 2.Patients who need endoscopic ultrasonography of pancreas; 3. Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Subjects who meet any of the following criteria cannot be selected for this trial:

First. The patient's physical condition does not meet the requirements of conventional endoscopic ultrasonography:

1. Poor physical condition, including hemoglobin ≤8.0g/dl, severe cardiopulmonary insufficiency, etc.
2. Anesthesia assessment failed
3. Pregnancy or breastfeeding
4. In the acute stage of chemical and corrosive injury, it is very easy to cause perforation
5. Recent acute coronary syndrome or clinically unstable ischemic heart attack
6. Heart disease patients with right-to-left shunt, patients with severe pulmonary hypertension (pulmonary artery pressure> 90mmHg),patients with uncontrolled systemic hypertension and patients with adult respiratory distress syndrome.

Second. Disagree to participate in this study.

Third. There are other problems that do not meet the requirements of this research or that affect the results of the research:

1. Pancreatic disease has undergone surgery or radiotherapy and chemotherapy beforehand;
2. Mental illness, drug addiction, inability to express themselves or other diseases that may affect follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 2 year
  The number of correctly classified images divided by the total number of images.
The completeness for standard station scanning | 2 year
  This was calculated as the number of stations successfully scanned divided by the total number of stations that should have been scanned.

SECONDARY OUTCOMES:
Cohen's kappa coefficient. | 2 year
  This data is to evaluate the agreement between the model and the endoscopists.
The completeness of anatomical landmarks | 2 year
  It calculated as the number of anatomical structures successfully scanned divided by the total number of structures that should have been scanned.
The completeness for standard stations and anatomical landmarks per individual | 2 year
  The completeness of stations and anatomic landmarks of biliopancreatic endoscopic ultrasonography by different endoscopists in the AI system assisted group and the control group were compared.
Operation time | 2 year
  In addition to puncture, elastography, and enhanced ultrasound to observe the lesion or treatment, it is also used to observe the time of biliopancreatic system.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, Doctor, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Some data underlying this trial cannot be shared publicly due to protection of participant's privacy.